CLINICAL TRIAL: NCT03251534
Title: Contribution of Stereography in the Quantification of Malunions Femoral Shaft Fractures Operated by Centromedullary Nailing. A Case Serie of 40 Patients
Brief Title: Contribution of Stereography (EOS Imaging System) in the Quantification of Femoral Shaft Fractures.
Acronym: FEOS
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: DCIC-1550
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Femoral Shaft Fracture
Keywords: Eos imaging stereography; Centromedullary nailing; Quantification of malunions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Centromedullary nailing

SUMMARY:
This observational study is a collection of clinical and imaging data of patients with a femoral shaft fracture treated by nails. The aim of this research is the contribution of the EOS imaging system in the quantification of malunions.

DETAILED DESCRIPTION:
The study is based on the collection of clinical and imaging data (using EOS imaging system) necessary for the follow-up of patients who have benefited, most often in the emergency, of a centromedullary nailing of the femoral shaft. The study does not lead to any further examination for the patient since they are followed until the removal of the material, which usually takes place 24 months after the fracture episode. This observational and pilot study is monocentric, prospective on a continuous series of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 16 years (parental agreement signed for minors) or adults at the time of data collection
* Patients with a femoral shaft fractures since january 2014
* Patients with a post-nailing femoral shaft fracture
* Patients with unilateral fracture
* Patients with regional origin allowing a follow-up in Grenoble center

Exclusion Criteria:

* Patients who refuse to sign a non-objective form
* Patients with femoral shaft fracture untreted with nails

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with surgery of femoral shaft fracture treated by nails
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Quantitative evaluation of rotational disturbances | 24 months
  Rotation disorder (degree angle), measured in a standardized and comparative way compared to the healthy side, by the EOS © software.

SECONDARY OUTCOMES:
Correlation of the rotation disorder with the clinical condition of the patient. | 24 months
  Rotation disorder (angle in degree).
Quantitative evaluation of the shortening or the lengthening of the operated limb (cranio-caudal plane). | 24 months
  Shortening or lengthening of the entire operative limb and of the femur alone (measured in mm), recorded in a standardized and comparative way compared to the healthy side, by the EOS © software
Correlation of shortening or limb lengthening with the clinical condition of the patient. | 24 months
  Shortening or lengthening of limb (measured in mm).
Quantitative evaluation of the varus-valgus (lateral-medial plane). | 24 months
  Varus-valgus (angle in degree), taken standardized and comparative way compared to the healthy side, by the EOS © software.
Correlation of the varus-valgus with the clinical condition of the patient | 24 months
  Varus-valgus (angle in degree).
Quantitative evaluation of the flessum-recurvatum | 24 months
  Flessum-recurvatum (angle in degree), measured in standardized and comparative way compared to the healthy side, by the EOS © software.
Correlation of the flessum-recurvatum with the clinical condition of the patient. | 24 months
  Flessum-recurvatum (angle in degree)
Idendification of the main risk factors of post-nailing rotational disturbances of femoral shaft fractures | 24 months
  Rotational disturbance (angle in degree)
Identification of the main risk factors of limb shortening or lengthening (cranio-caudal plane) after femoral nailing of femoral shaft fractures. | 24 months
  Shortening or limb lengthening (measured in mm).
Identification of the main risk factors for the varus-valgus (lateral-medial plane) after femoral nailing of fhe femoral shaft fractures | 24 months
  Varus-valgus (angle in degree).
Identification of the main risk factors of the flessum-recurvatum after femoral nailing of fhe femoral shaft fractures | 24 months
  Flessum-recurvatum (angle in degree).

CONTACTS AND LOCATIONS:
Overall Officials: Tonetti Jerôme, MD, PhD, Principal Investigator — Orthopedic and Trauma department, University Hospital, Grenoble
Locations (1):
- Orthopedic and Trauma Department, University Hospital, Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Investigation Centre for Innovative Technology Network — http://www.cic-it.fr/cic-it-grenoble.php